CLINICAL TRIAL: NCT01588054
Title: Prospective Radiographic and Clinical Evaluation of Surgical Treatment for Cervical Deformity: A Multi-Center Study
Brief Title: Prospective Radiographic and Clinical Evaluation of Surgical Treatment for Cervical Deformity
Acronym: PCD
Status: Completed | Type: Observational
Sponsor: International Spine Study Group Foundation (Other)
Collaborators: DePuy Spine (Industry)
Responsible Party: Sponsor
Other Study IDs: 2107-01
Record Dates: First submitted 2012-04-24; First posted 2012-04-30 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Cervical Deformity; Kyphosis; Scoliosis
MeSH Terms: conditions — Kyphosis; Scoliosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- adults, cervical deformity, surgical treatment: Adults 18years or older at time of enrollment, cervical deformity to include kyphosis (C2-7 greater than 10 degrees) or scoliosis (coronal cobb greater than 10 degrees), plans for surgical treatment of cervical deformity

SUMMARY:
The purpose of this study is to define clinical and demographic features within the population suffering from cervical deformity to assist health professionals to make important treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years of age or greater
* Cervical deformity (kyphosis C2-7 greater than 10 degrees or scoliosis with coronal cobb greater than 10 degrees)
* Plans for surgical correction of cervical deformity

Exclusion Criteria:

* Active tumor or infection
* Acute trauma
* Unwillingness to provide consent or complete study forms
* Prisoner
* Pregnant or planning to get pregnant during study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: spine surgeon clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-01-09 (Actual); Primary Completion 2021-05-08 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Radiographs | Prior to surgery, 8-16 weeks postop, 4-8 months postop, 9-23 months postop, and 24-30 months postop
  Changes in the degree of deformity post surgical correction and assessment of fusion.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | Prior to surgery, 8-16 weeks postop, 4-8 months postop, 9-23 months postop, and 24-30 months postop
  Changes related to worsening/improved neck pain as regards ability to manage everyday life.
Numeric rating scale (NRS) | Prior to surgery, 8-16 weeks postop, 4-8 months postop, 9-23 months postop, and 24-30 months postop
  Changes in level of neck and back pain within the past month
CSRS SWAL-QOL | Prior to surgery, 8-16 weeks postop, 4-8 months postop, 9-23 months postop, and 24-30 months postop
  Changes with swallowing problems affecting day-to-day quality of life
EQ-5D3L | Prior to surgery, 8-16 weeks postop, 4-8 months postop, 9-23 months postop, and 24-30 months postop
  Changes in current health state
mJOA | Prior to surgery, 8-16 weeks postop, 4-8 months postop, 9-23 months postop, and 24-30 months postop
  Changes in neck pain regarding ability fo function in everyday life

CONTACTS AND LOCATIONS:
Overall Officials: Justin Smith, MD, PhD, Principal Investigator
Locations (10):
- United States (10):
  - Scripps Clinic La Jolla, La Jolla, California
  - University of California - Davis, Sacramento, California
  - University of California - San Francisco Medical Center, San Francisco, California
  - Denver International Spine Center, Denver, Colorado
  - University of Kansas Medical Center, Kansas City, Kansas
  - Washington University, St Louis, Missouri
  - New York University - Hospital for Joint Diseases, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Baylor Scoliosis Center, Plano, Texas
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Smith JS, Ben-Israel D, Kelly MP, Lafage V, Lafage R, Klineberg EO, Kim HJ, Line B, Protopsaltis TS, Passias P, Eastlack RK, Mundis GM, Riew KD, Kebaish K, Park P, Gupta MC, Gum JL, Daniels AH, Diebo BG, Hostin R, Scheer JK, Soroceanu A, Hamilton DK, Buell TJ, Lewis SJ, Lenke LG, Mullin JP, Schwab FJ, Burton D, Shaffrey CI, Ames CP, Bess S. The gap between surgeon goal and achieved sagittal alignment in adult cervical spine deformity surgery. J Neurosurg Spine. 2025 Jan 3;42(3):309-319. doi: 10.3171/2024.8.SPINE24703. Print 2025 Mar 1. PMID 39752660